CLINICAL TRIAL: NCT07085065
Title: Virtual Reality to Reduce Pain and Anxiety in Hematological Cancer Patients Undergoing Invasive Procedures: Protocol for a Crossover Clinical Trial
Brief Title: Distraction With Virtual Reality From Pain and Anxiety for Patients With Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yesmine Amara (Other)
Collaborators: University of Sfax (Other)
Responsible Party: Sponsor-Investigator, Yesmine Amara, Principal Investigator-PhD student, University of Sfax
Organization: University of Sfax (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMS-2025-VR1024
Record Dates: First submitted 2025-07-10; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Anxiety; Procedures; Hematological Neoplasms
Keywords: Virtual Reality; Pain; Anxiety; Hematological Malignancies; Invasive procedures; Chemotherapy
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Hematologic Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: The intervention consists of a complete sequence involving three phases: Period 1 (standard care), a washout period of at least seven days, and Period 2 (VR session). In addition to this internal control design, the study will also include an external control group consisting of patients who will receive only standard care throughout the study. These external control participants will be matched to the interventional group based on age and procedure type, ensuring comparability between groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal control design (Experimental): The intervention consists of a complete sequence involving three phases: Period 1 (standard care), a washout period of at least seven days, and Period 2 (VR session during the same procedure).
  Interventions: Device: VR session
- external control group (Active Comparator): This arm consists of patients who will receive only standard care throughout the study. These external control participants will be matched to the interventional group based on age and procedure type, ensuring comparability between groups.
  Interventions: Device: VR session

INTERVENTIONS:
Device: VR session — Standard care: Standard care. In both the external control group and the intervention group during Period 1, painful procedures will be performed ccording to usual clinical practice by trained healthcare professionals.
  VR session: The device includes a VR headset connected to a smartphone, which displays immersive visual content, along with headphones that deliver audio content. Scenarios are culturally and demographically adapted to the study population. The duration of each VR session will correspond to the time required for each painful procedure.
  Other Names: Standard care

SUMMARY:
The goal of this clinical trial] is to study the effectiveness of Virtual Reality (VR) in reducing pain and anxiety during painful procedures for patients with hematological malignancies The main question[s] it aims to answer are:

Does VR effectively reduce pain during painful procedures for patients with hematological malignancies ? Does VR effectively reduce anxiety during painful procedures for patients with hematological malignancies ? Interventional group (intra-group comparaison): This design allows each patient to act as his own control.: The intervention consists of a complete sequence involving three phases: Period 1 (standard care), a washout period of at least seven days, and Period 2 (VR session).

External control group (inter-group comparaison): Patients will be assigned to the intervention group first, and then a matching external control patient will be selected based on age and type of procedure.

DETAILED DESCRIPTION:
This study is a prospective interventional crossover trial designed to evaluate the efficacy of Virtual Reality during painful procedures, including Bone Marrow Biopsy, Bone Marrow Aspiration, Lumbar Puncture, Venipuncture, and chemotherapy. Previous studies have suggested that virtual reality (VR) can distract patients from painful stimuli, enhance the quality of healthcare, and improve overall patient well-being.

ELIGIBILITY:
Inclusion Criteria

* being ≥ 6 years old
* having a confirmed diagnosis of a hematological malignancy
* undergoing at least one of the following procedures: Bone Marrow Biopsy, Bone Marrow Aspiration, Lumbar Puncture, Venipuncture, or Chemotherapy.

Exclusion Criteria:

* unstable or photosensitive epilepsy
* hearing, visual, or inner ear impairments
* severe psychiatric, cognitive, or mental disorders
* Contagious diseases
* Communication difficulties
* Patients who withdraw consent
* Patient who remove the VR headset during the procedure

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain levels using the Numeric Rating Scale (0-10) | Assessed within 5 minutes before the procedure and within 5 minutes after the procedure
  The Numeric rating scale (NRS) of pain is a scale from 0 to 10, where scores from 0 to 3 indicate mild pain, 4 to 6 indicate moderate pain, and 7 to 10 indicate severe pain. The NRS has been proven valid and reliable for measuring cancer-related pain. It will be assessed within 5 minutes before the procedure and within 5 minutes after the procedure during the two periods (standard care, VR session)

SECONDARY OUTCOMES:
Change in Anxiety using the Spielberger State-Trait Anxiety Inventory (Y1 and Y2) | Trait anxiety: Baseline State anxiety: Assessed within 5 minutes before the procedure and within 5 minutes after the procedure
  The Spielberger Trait Anxiety Inventory measures an individual's general tendency to experience anxiety across various situations. This inventory reflects a stable personality trait, meaning some individuals are more prone to anxiety than others. It will be measured at Baseline The Spielberger State Anxiety Inventory assesses anxiety as a temporary emotional state or condition triggered by a specific situation or stimulus. This scale measures "here and now" anxiety, which can fluctuate in intensity. The STAI-Y1 consists of 20 items, with scores ranging from 20 to 80, evaluated on a 4-point Likert scale (ranging from "Not at all" to "Completely"). Higher scores on both subscales indicate higher levels of anxiety. It will be assessed within 5 minutes before the procedure and within 5 minutes after the procedure during the two periods (standard care and VR session)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical hematology department of unversity hospital of Hedi Chaker of Sfax, Tunisia, Tunis, Sfax Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No